CLINICAL TRIAL: NCT01272258
Title: A Phase 2b, Randomized, Double-Blind, Placebo-Controlled Clinical Trial of Observed Systemic, Long-Acting, Anti-HIV Treatment With a Monoclonal Anti CCR5 Antibody (PRO 140) as an Adjunct to a New, Optimized, Oral Antiretroviral Regimen in HIV-Infected Injection Drug Users With Viral Rebound and Documented Poor Adherence to the Previous Antiretroviral Regimen
Brief Title: A Trial of Observed Long-acting, Anti-HIV Treatment With a Monoclonal CCR5 Antibody (PRO 140) as an Adjunct to a New, Optimized, Oral Antiretroviral Regimen in HIV-infected Injection Drug Users With Viral Rebound and Documented Poor Adherence
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: CytoDyn, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRO 140 2102
Record Dates: First submitted 2011-01-05; First posted 2011-01-07 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-01

CONDITIONS: HIV
MeSH Terms: interventions — leronlimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): PRO 140
  Interventions: Drug: PRO 140
- Arm 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PRO 140 — SC injection
  Arms: Arm 1
Drug: Placebo — SC injection
  Arms: Arm 2

SUMMARY:
PRO 140 2102 is a phase 2b, national, multicenter, randomized, double-blind, placebo-controlled study in order to evaluate the safety and efficacy of PRO 140 (anti-CCR5 monoclonal antibody) administered subcutaneously as an adjunct to a new, optimized, oral antiretroviral regimen in HIV-infected injection drug users with viral rebound and documented poor adherence to the previous antiretroviral regimen.

ELIGIBILITY:
Key Inclusion Criteria:

1. Only R5 virus
2. HIV-1 RNA > 1,000 copies/mL but < 100,000 copies/mL
3. CD4+ lymphocyte counts > 100 cells/μL
4. Non-prescription recreational drug use within the previous 6 months

Key Exclusion Criteria:

1. Females who are pregnant (positive blood test), lactating, or breastfeeding, or who plan to become pregnant during the study
2. Prior use of any CCR5 entry inhibitors
3. History of any acquired immune deficiency syndrome (AIDS)-defining illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-12; Primary Completion 2017-01 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Specific measure that will be used to determine the effect of the interventions: Percentage of subjects without virologic failure at week 24. | 24 Weeks
  Percentage of subjects without virologic failure at week 24.

CONTACTS AND LOCATIONS:
Locations (1):
- Drexel University College of Medicine, Philadelphia, Pennsylvania, United States